CLINICAL TRIAL: NCT03497975
Title: A Phase 2b/3, Randomized, Double-Blind, Placebo-Controlled, 2-Arm, Efficacy and Safety Study in Prurigo Nodularis (PN) With Nalbuphine ER Tablets for Pruritus Relief Through Itch Scratch Modulation (PRISM Study)
Brief Title: PRISM Study-Pruritus Relief Through Itch Scratch Modulation
Acronym: PRISM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Trevi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TR11; 2018-001219-53 (EudraCT Number)
Record Dates: First submitted 2018-03-22; First posted 2018-04-13 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Prurigo Nodularis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NAL ER (Experimental): During the double-blind (DB) period, participants were titrated over 2 weeks to NAL ER 162 mg, orally, twice daily (BID), followed by 162 mg, orally, BID, for 12 weeks. During the open label extension (OLE) period, participants perceived a titration period of 2 weeks, and continued to receive NAL ER 162 mg, orally, BID, for 38 weeks in total.
  Interventions: Drug: Nalbuphine ER Tablets
- Placebo (Placebo Comparator): During the DB period, participants perceived a titration period of 2 weeks during which they received placebo to match the active titration period, followed by placebo, orally, BID, for 12 weeks. During the OLE period, participants were titrated over 2 weeks to NAL ER 162 mg, orally, BID, which they received for 38 weeks (including titration).
  Interventions: Drug: Nalbuphine ER Tablets; Drug: Placebo Tablets

INTERVENTIONS:
Drug: Nalbuphine ER Tablets — Active Nalbuphine ER Tablets
  Other Names: NAL ER Tablets
Drug: Placebo Tablets — Placebo matching NAL ER with no active substance
  Arms: Placebo

SUMMARY:
To investigate the anti-pruritic efficacy and safety of Nalbuphine Extended Release (ER) (NAL ER) tablets in Prurigo Nodularis. Participants were randomized to NAL ER (or matching placebo) with the primary endpoint evaluation at Week 14. During the open label extension, participants who received NAL ER were continued on NAL ER and participants who received placebo would then shift to NALER.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with generalized nodular PN, covering 2 separate body parts, and 10 or more pruriginous nodules
* Severe itch due to PN
* Age 18 years and older at the time of consent, and a life expectancy of at least 18 months.
* Individuals using antidepressants must be on a stable dose for a minimum of 4 weeks prior to screening.
* Participants with a history of acute secondary dermatoses within the preceding 6 months may enroll only if the dermatosis has resolved completely as follows per medical history or participant self-report and current clinical assessment: (a) Localized contact dermatitis, environmental exposures, superficial burns, or viral exanthems must have been resolved for at least 4 weeks prior to screening. (b) Skin or environmental infestations, such as scabies, lice, or bed bugs, must have been resolved for at least 8 weeks prior to screening.
* Any identified systemic, non-dermatologic disease that could be a potential cause of concomitant pruritus (e.g., thyroid disease, celiac disease, hepatitis C virus [HCV]) must either have resolved, been successfully treated [i.e., HCV ribonucleic acid (RNA) negative], or must be successfully managed with stable, optimized treatment (e.g., thyroid replacement, dietary management with resolution of symptoms, respectively) for at least 3 months prior to screening.
* Participants who are human immunodeficiency virus (HIV) positive may enroll if they meet the following criteria: (a) currently on a stable (> 6 months stable use) and well tolerated highly active antiretroviral therapy regimen; (b) cluster of differentiation 4 (CD4) count > 500 cells/mL; and (c) HIV ribonucleic acid (RNA) < 50 copies/mL documented for at least 6 months prior to enrollment.

Exclusion Criteria:

* Pruritus due to localized PN (only one body part affected), or less than 10 nodules
* Active, uncontrolled, pruritic dermatoses in need of treatment (such as atopic dermatitis or bullous pemphigoid for example).
* History of a major psychiatric disorder such as bipolar disorder or schizophrenia. History of active substance abuse in the last 3 years.
* Known intolerance [gastrointestinal (GI), central nervous system (CNS) symptoms] or hypersensitivity/drug allergy to opioids.
* Use of certain concomitant medications and treatments within a period prior to the study, or requirement for these medications during the study:

  * Potential participants taking opiates, gabapentin, pregabalin, calcineurin inhibitors, cannabinoid agonists, capsaicin, cryosurgery, topical doxepin, thalidomide or methotrexate, topical antihistamines or topical corticosteroids require a 14-day washout.
  * Within 4 weeks prior to screening: ultraviolet (UV)-therapy, exposure to any investigational medication, including placebo
  * Within 3 months prior to screening: Non-insulin biologics (including monoclonal antibodies) that modify the immune system,
  * Individuals taking monoamine oxidase inhibitors are excluded, as concomitant opiate use may increase the risk for serotonin syndrome.
* Myocardial infarction or acute coronary syndrome within the previous 3 months, as reported by the participant.
* Individuals with prolonged QT interval corrected for heart rate using Fridericia's formula (QTcF).

Note: Other Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2023-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Development Officer, Study Director — Trevi Therapeutics
Locations (70):
- United States (36):
  - Study Site 151, Phoenix, Arizona
  - Study Site 121, Fremont, California
  - Study Site 157, Laguna Niguel, California
  - Study Site 141, North Hollywood, California
  - Study Site 130, San Francisco, California
  - Study Site 128, Washington D.C., District of Columbia
  - Study Site 138, Boca Raton, Florida
  - Study Site 158, Orlando, Florida
  - Study Site 108, South Miami, Florida
  - Study Site 142, Tampa, Florida
  - Study Site 102, Rockville, Maryland
  - Study Site 136, Boston, Massachusetts
  - Study Site 153, Brighton, Massachusetts
  - Study Site 143, Ann Arbor, Michigan
  - Study Site 139, Troy, Michigan
  - Study Site 118, Saint Joseph, Missouri
  - Study Site 144, Henderson, Nevada
  - Study Site 146, Las Vegas, Nevada
  - Study Site 109, Portsmouth, New Hampshire
  - Study Site 159, Hackensack, New Jersey
  - Study Site 134, Stony Brook, New York
  - Study Site 101, Wilmington, North Carolina
  - Study Site 122, Cincinnati, Ohio
  - Study Site 120, Cleveland, Ohio
  - Study Site 132, Hershey, Pennsylvania
  - Study Site 106, Philadelphia, Pennsylvania
  - Study Site 131, Johnston, Rhode Island
  - Study Site 147, Charleston, South Carolina
  - Study Site 107, Charleston, South Carolina
  - Study Site 140, Chattanooga, Tennessee
  - Study Site 145, Knoxville, Tennessee
  - Study Site 137, Austin, Texas
  - Study Site 103, Webster, Texas
  - Study Site 150, West Jordan, Utah
  - Study Site 135, Spokane, Washington
  - Study Site 148, Morgantown, West Virginia
- Austria (2):
  - Study Site 401, Graz
  - Study Site 402, Linz
- France (2):
  - Study Site 501, Brest
  - Study Site 502, Paris
- Germany (16):
  - Study Site 204, Frankfurt am Main, Hesse
  - Study Site 202, Münster, North Rhine-Westphal
  - Study Site 201, Mainz, Rhineland-Palatinate
  - Study Site 213, Dresden, Saxony
  - Study Site 205, Bad Bentheim
  - Study Site 216, Berlin
  - Study Site 209, Berlin
  - Study Site 208, Berlin
  - Study Site 219, Cologne
  - Study Site 221, Düsseldorf
  - Study Site 215, Hamburg
  - Study Site 222, Hamburg
  - Study Site 212, Heidelberg
  - Study Site 214, Kiel
  - Study Site 220, München
  - Study Site 206, Stuttgart
- Poland (14):
  - Study Site 304, Bialystok
  - Study Site 306, Katowice
  - Study Site 308, Krakow
  - Study Site 316, Krakow
  - Study Site 309, Lodz
  - Study Site 314, Lublin
  - Study Site 305, Ostrowiec Świętokrzyski
  - Study Site 313, Poznan
  - Study Site 315, Poznan
  - Study Site 303, Rzeszów
  - Study Site 310, Warsaw
  - Study Site 301, Warsaw
  - Study Site 312, Warsaw
  - Study Site 302, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 70 sites in Germany, Poland, Austria, France and the United States from 07 August 2018 to 24 February 2023.
Pre-assignment Details: A total of 608 participants were screened, out of which 353 participants were randomized, and 344 participants were treated with NAL ER and/or placebo.
Period: Overall Study
Arm/Group | NAL ER | Placebo
Started | 173 | 180
Modified Intent-to-treat (mITT) Analysis Set (The mITT population included all randomized participants who received at least a single dose of investigational product (IP).) | 168 | 176
Participants Who Entered the OLE Period | 107 | 144
Completed | 71 | 80
Not Completed | 102 | 100
Not completed — Withdrew Consent | 34 | 35
Not completed — Lost to Follow-up | 7 | 7
Not completed — Physician Decision | 4 | 5
Not completed — Discontinued | 42 | 39
Not completed — Reason Not Specified | 15 | 14

BASELINE CHARACTERISTICS:
Population: The mITT population included all randomized participants who received at least a single dose of IP.
Groups:
- NAL ER: During the DB period, participants were titrated over 2 weeks to NAL ER 162 mg, orally, BID, followed by 162 mg, orally, BID, for 12 weeks. During the OLE period, participants perceived a titration period of 2 weeks, and continued to receive NAL ER 162 mg, orally, BID, for 38 weeks in total.
- Total: Total of all reporting groups
Arm/Group | NAL ER | Placebo | Total
Number analyzed (Participants) | 168 | 176 | 344
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (13.25) | 55.9 (14.32) | 57.7 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 112 | 212
  Male | 68 | 64 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 63 | 66 | 129
  Unknown or Not Reported | 99 | 103 | 202
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 6 | 11 | 17
  Black or African American | 24 | 23 | 47
  White | 132 | 134 | 266
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Worst Itch - Numerical Rating Scale (WI-NRS) Score [Mean (Standard Deviation); unit: score on scale] — Population: NRS is a patient related outcome (PRO) instrument to quantify the intensity of worst itching experienced for 24-hour period and can be applied and validated either with reference to the average itch or to the absolute worst itch (WI-NRS). WI-NRS is a set of boxes, one for each number, from 0 (no itching) to 10 (worst possible itching). Higher scores indicate worst itching experience. "Number analyzed" indicates number of participants with data available for analysis at a specified timepoint.
  score on scale
    number analyzed (Participants) | 167 | 176 | 343
    (all) | 8.637 (0.9115) | 8.650 (0.8902) | 8.643 (0.8993)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥ 4- Point Decrease in 7-day Average Worst Itch - Numerical Rating Scale (WI-NRS) up to Week 14
Description: The NRS is a patient related outcome (PRO) instrument, designed to quantify the intensity of worst itching experienced during a 24-hour period, and can be applied and validated either with reference to the average itch or to the absolute worst itch (WI-NRS) over that 24-hour period. WI-NRS is a set of boxes, one for each number, from 0 (no itching) to 10 (worst possible itching). Higher scores indicate worst itching experience. Responder was defined as a participant with a ≥4-point decrease in the 7-day average WI-NRS from baseline to Week 14.
Time Frame: Baseline up to Week 14
Population: The mITT population included all randomized participants who received at least a single dose of IP. Overall number of participants analyzed indicates number of participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 99 | 131
percentage of participants | 24.24 | 14.50
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Test type: Superiority; p = 0.0309, Regression, Logistic — Logistic regression model includes WI-NRS baseline score as a covariate, treatment and the study site (with pooling) as a fixed effect; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.07 to 4.13]

2. Secondary Outcome: Change From Baseline in Itch-related Quality of Life (ItchyQoL) Total Score at Week 14
Description: The ItchyQoL consists of 22 pruritus-specific items measuring how pruritus affects participant's QoL in the area of symptoms related to the itch condition (6 questions), functional limitations (7 questions), and emotions (9 questions). The participant scored each question never = 1, rarely = 2, sometimes = 3, often = 4, all the time = 5. The ItchyQoL total score were obtained as the sum of the 22 items ranging from 22 to 110, with higher score indicating worsening of pruritus. A negative change from baseline indicated improvement in the pruritus-related difficulties.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 95 | 127
score on a scale | -17.4 (18.01) | -8.8 (17.15)
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Test type: Superiority; p = 0.0002, Mixed Model for Repeated Measurements — Repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline ItchyQoL value. An unstructured covariance matrix is used; Difference in LS Mean = -7.06, 95% CI 2-sided [-10.82 to -3.30], Standard Error of Mean 1.91

3. Secondary Outcome: Change From Baseline in Prurigo Activity Score (PAS) Assessed by the Percentage of Participants With 1-Category Improvement in the Percentage of Pruriginous Lesions With Excoriations/Crusts (Item 5a) at Week 14
Description: PAS consists of 5 quantitative/qualitative measurements related to examination of skin: Type; number;distribution;quantitative number of lesions in a body part;activity. Prurigo lesion activity is recorded as a stage (0 to 4), based on percentage of overall lesions with relevant characteristic. Three types of PAS responders defined one for each of the following items: Pruriginous lesions with excoriations/crusts (item 5a);Healed lesions (item 5b);Number of lesions (item 2). Pruriginous lesions with excoriations/crusts (item 5a) was recorded from 0 to 4;where 0 = 0-25%1 = 26-50%,2 = 51-75%,3 = 76-90%,4 = 91-100%. Higher score=a greater number of pruriginous lesions with excoriations/crusts. A responder was defined as a participant who has at least 1-category improvement in the relevant item from baseline to Week 14. Baseline is defined as the last non-missing evaluation (including repeated and unscheduled assessments) taken prior to or on the date of first dose of study medication.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 112 | 146
percentage of participants | 54.5 | 41.1
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Test type: Superiority; p = 0.0179, Regression, Logistic — Logistic regression model includes PAS (Item 5a) baseline score as a covariate, treatment as a fixed effect and the study site (with pooling) as a fixed effect; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.11 to 3.07]

4. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 8a at Week 14
Description: PROMIS Sleep Disturbance Short Form 8a questionnaire is a tool for assessing sleep. It has 8 questions which measures sleep in the past 7 days.There is 1 broad sleep quality question with options:"very poor","poor","fair","good",and "very good".Remaining 7 questions are answered with:"not at all","a little bit","somewhat","quite a bit",and "very much".Lowest possible raw score=8; highest possible raw score=40. The T-score rescales raw score into a standardized score with a mean of 50 and an standard deviation of 10 derived from general population.Lowest possible T-score=28.9;highest possible T-score=76.6.Higher T-score shows more of the concept measured,higher the T-Score worse the sleep disturbance.Scores <55=normal limits, 55-60=mild, 61-70=moderate,and >70=severe sleep disturbance.Baseline=last non-missing evaluation (including repeated and unscheduled assessments) taken prior to or on the date of first dose of study medication.Negative change from baseline indicated better sleep.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 96 | 127
T-score | -9.5 (10.01) | -4.5 (8.44)
Statistical Analysis 1: Comparison: NAL ER vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measurements — Repeated measures model with the fixed effects of treatment, visit, treatment by visit interaction and baseline PROMIS value. An unstructured covariance matrix is used; Difference in LS Mean = -4.43, 95% CI 2-sided [-6.55 to -2.31], Standard Error of Mean 1.08

5. Secondary Outcome: Change From Baseline in 7-Day Average WI-NRS to Week 14
Description: The NRS is a PRO instrument, designed to quantify the intensity of worst itching experienced during a 24-hour period, and can be applied and validated either with reference to the average itch or to the absolute worst itch (WI-NRS) over that 24-hour period. WI-NRS is a set of boxes, one for each number, from 0 (no itching) to 10 (worst possible itching). Higher scores indicate worst itching experience. Baseline WI-NRS value was calculated as the arithmetic mean of the WI-NRS values (minimum of 5 required) taken for eligibility review by site at the time of randomization. A negative change from baseline indicates improvement in symptoms.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 99 | 131
score on a scale | -2.5 (2.36) | -1.6 (2.14)

6. Secondary Outcome: Change From Baseline in PAS Assessed by the Percentage of Participants With 1-Category Improvement in the Percentage of Healed Lesions (Item 5b) at Week 14
Description: PAS consists of 5 quantitative/qualitative measurements related to skin-Type; number; distribution; quantitative number of lesions in body part; activity. Prurigo lesion activity is recorded as stage (0 to 4), based on percentage of overall lesions with relevant characteristic. Three types of PAS responders are defined: Pruriginous lesions with excoriations/crusts (item 5a); Healed lesions (item 5b); Number of lesions (item 2). Prurigo lesions (item 5b), where 0 = 100%,1 = 75-99%,2 = 50-74%,3 = 25-49%,4 = 0-24% healed pruriginous lesions. Lower score=more number of healed pruriginous lesions. A responder was defined as a participant who has at least 1-category improvement in the relevant item from baseline to Week 14. Baseline was defined as the last non-missing evaluation (including repeated and unscheduled assessments) taken prior to or on the date of first dose of treatment. A negative change from baseline would indicate higher number of healed lesions.
Time Frame: Baseline, Week 14
Population: The mITT population included all randomized participants who received at least a single dose of IP.
Measure: Number; unit: percentage of participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 168 | 176
percentage of participants | 39.3 | 34.7

7. Secondary Outcome: Change From Baseline in PAS Assessed by the Percentage of Participants With 1-Category Improvement in the Percentage of Lesions (Item 2) at Week 14
Description: PAS consists of 5 quantitative/qualitative measurements of skin- Type; number; distribution; quantitative number of lesions in body part; activity. Prurigo lesion activity is recorded as stage (0 to 4) based on percentage of overall lesions with relevant characteristic. Three types of PAS responders are defined: Pruriginous lesions with excoriations/crusts (item 5a); Healed lesions (item 5b); Number of lesions (item 2). Prurigo lesion activity is recorded as a stage (0 to 4), based on the percentage of overall lesions with the relevant characteristic. A lower score indicates less number of pruriginous lesions. A responder was defined as a participant who has at least 1-category improvement in the relevant item from baseline to Week 14. Baseline was defined as the last non-missing evaluation (including repeated and unscheduled assessments) taken prior to or on the date of first dose of study medication. A negative change from baseline would indicate lower number of lesions.
Time Frame: Baseline, Week 14
Population: The mITT population included all randomized participants who received at least a single dose of IP.
Measure: Number; unit: percentage of participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 168 | 176
percentage of participants | 25.0 | 18.8

8. Secondary Outcome: Change From Baseline in Investigator Global Assessment-Prurigo Nodularis (IGA-PN) Assessed by the Percentage of Participants With 1-Category Improvement in Activity at Week 14
Description: The IGA-PN collects an investigator global assessment of status of PN skin lesions. The IGA-PN uses a 5-category scale (scoring 0 to 4) to describe the status of 2 aspects of disease: The Activity (amount of excoriation and crusting associated with the prurigo lesions), and the Stage (the quantitative presence and proportion of flattening of the lesions). The excoriation/crusting activity on the surface (PN-Activity) where it considers number of PN lesion with excoriations and crusts on the top, 0=clear (No nodules), 1 =small number, 2=minority of nodules, 3=most nodules, 4=severe (vast majority of nodules). A higher number indicates severe status of PN skin lesions. An IGA-PN responder for activity was defined as participants who has at a least 1-category improvement in the respective score from baseline to Week 14. Baseline was defined as the last non-missing evaluation (including repeated and unscheduled assessments) taken prior to or on the date of first dose of study medication.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 112 | 146
percentage of participants | 57.1 | 41.1

9. Secondary Outcome: Change From Baseline in IGA-PN Assessed by the Percentage of Participants With 1-Category Improvement in Stage at Week 14
Description: The IGA-PN collects an investigator global assessment of status of PN skin lesions. The IGA-PN uses a 5-category scale(scoring 0 to 4) to describe 2 aspects of disease. The Activity(amount of excoriation and crusting of prurigo lesions) and the Stage(the quantitative presence and proportion of flattening of lesions),where 0=clear(No nodules),1=Rare, flattened lesions, with no more than single dome-shaped palpable nodules(1-5 nodules), 2=Few,mostly flattened lesions, with small number of dome-shaped palpable nodules(6-19 nodules,3=Many lesions, partially flattened and dome-shaped palpable nodules (20-100 nodules),4=Abundant lesions, majority are dome-shaped palpable nodules (over 100 nodules).Higher number= presence of abundant lesions.Responder as defined as participants who has at a least 1-category improvement from baseline to Week 14.Baseline was defined as the last non-missing evaluation(repeated and unscheduled assessments)taken prior to or on the date of first dose of treatment.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 112 | 146
percentage of participants | 43.8 | 32.9

10. Secondary Outcome: Percentage of Participants Having a Patient Benefit Index, Pruritus Version (PBI-P) Score of ≥1 at Week 14
Description: PBI-P is an instrument that measures participant-defined treatment objectives and benefits acquired during the course of treatment.During and after therapy, the participant completes a matched "on-treatment" Treatment Benefits questionnaire and rates the extent to which the treatment objectives have been achieved.It consists of 27 multiple choice questions that can be answered "not at all","somewhat","moderately","quite","very".PBI-P global score is computed according to the score obtained for patient needs questionnaire (PNQ) and patient benefit questionnaire (PBQ).Score may only be computed if the participant has provided valid data on importance (PNQ) and benefit (PBQ) for at least 75% of the respective treatment goals,i.e., for at least 21 of the 27 items. Total score ranges from 0-135. Higher scores=more benefit received from the study to the participant.Responses "does/did not apply","question answered" are considered valid values when counting number of non-missing responses.
Time Frame: At Week 14
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 87 | 95
percentage of participants | 100.0 | 100.0

11. Secondary Outcome: Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, and Discontinued From Study Drug Due to TEAEs in DB Period
Description: An AE is any untoward medical occurrence in a participant who administered a pharmaceutical product, and which does not necessarily have to have a causal relationship with the study drug. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. DB period TEAEs are defined as AEs that either start or worsen in severity on or after the first DB dose and prior to the first extension titration dose of study medication in the OLE period. TEAEs included both serious & non-serious TEAEs.
Time Frame: Baseline up to Week 14
Population: The safety population included all randomized participants who received at least a single dose of IP.
Measure: Count of Participants; unit: Participants
Groups:
- NAL ER: During the DB period, participants were titrated over 2 weeks to NAL ER 162 mg, orally, BID, followed by 162 mg, orally, BID, for 12 weeks.
- Placebo: During the DB period, participants perceived a titration period of 2 weeks during which they received placebo to match the active titration period, followed by placebo, orally, BID, for 12 weeks.
Arm/Group | NAL ER | Placebo
Number analyzed (Participants) | 168 | 176
Participants
  Participants with TEAEs | 136 | 106
  Participants with Serious TEAEs | 9 | 8
  Participants with Study Drug Discontinuation Due to TEAEs | 53 | 13

12. Secondary Outcome: Number of Participants Who Experienced TEAEs, Serious TEAEs, and Discontinued From Study Drug Due to TEAEs in OLE Period
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the study drug. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. OLE period TEAEs are defined as AEs that either start or worsen in severity on or after the first extension titration dose of study medication. TEAEs included both serious & non-serious TEAEs.
Time Frame: From Week 14 up to Week 56
Population: The safety population included all randomized participants who received at least a single dose of IP. Overall number of participants analyzed indicates number of participants who entered OLE period.
Measure: Count of Participants; unit: Participants
Groups:
- Prior NAL ER (OLE Period): During the OLE period, participants perceived a titration period of 2 weeks, and continued to receive NAL ER 162 mg, orally, BID, for 38 weeks in total.
- Prior Placebo (OLE Period): During the OLE period, participants were titrated over 2 weeks to NAL ER 162 mg, orally, BID, which they received for 38 weeks (including titration).
Arm/Group | Prior NAL ER (OLE Period) | Prior Placebo (OLE Period)
Number analyzed (Participants) | 107 | 144
Participants
  Participants with TEAEs | 84 | 116
  Participants with Serious TEAEs | 7 | 7
  Participants with Study Drug Discontinuation Due to TEAEs | 8 | 30

ADVERSE EVENTS:
Time Frame: DB Period: Baseline up to Week 14; OLE Period: From Week 14 to Week 56
Description: The safety population included all randomized participants who received at least a single dose of IP.
Groups:
- NAL ER (DB Period): During the DB period, participants were titrated over 2 weeks to NAL ER 162 mg, orally, BID, followed by 162 mg, orally, BID, for 12 weeks.
- Placebo (DB Period): During the DB period, participants perceived a titration period of 2 weeks during which they received placebo to match the active titration period, followed by placebo, orally, BID, for 12 weeks.
Arm/Group | NAL ER (DB Period) | Placebo (DB Period) | Prior NAL ER (OLE Period) | Prior Placebo (OLE Period)
All-Cause Mortality (participants affected / at risk) | 0/168 | 0/176 | 0/107 | 0/144
Serious Adverse Events (participants affected / at risk) | 9/168 | 8/176 | 7/107 | 7/144
Other Adverse Events (participants affected / at risk) | 112/168 | 58/176 | 49/107 | 95/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NAL ER (DB Period) (N=168) | Placebo (DB Period) (N=176) | Prior NAL ER (OLE Period) (N=107) | Prior Placebo (OLE Period) (N=144)
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 0 | 1
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Serous cystadenocarcinoma ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1
Dissociation (Psychiatric disorders) | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NAL ER (DB Period) (N=168) | Placebo (DB Period) (N=176) | Prior NAL ER (OLE Period) (N=107) | Prior Placebo (OLE Period) (N=144)
Nausea (Gastrointestinal disorders) | 52 | 16 | 13 | 44
Constipation (Gastrointestinal disorders) | 26 | 7 | 4 | 11
Vomiting (Gastrointestinal disorders) | 19 | 6 | 3 | 20
Dizziness (Nervous system disorders) | 53 | 6 | 5 | 30
Headache (Nervous system disorders) | 26 | 14 | 8 | 22
Somnolence (Nervous system disorders) | 25 | 6 | 3 | 19
Fatigue (General disorders) | 23 | 10 | 5 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 9 | 5 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 0 | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 10 | 15
Treatment noncompliance (General disorders) | 4 | 3 | 8 | 8
Medication error (Injury, poisoning and procedural complications) | 4 | 6 | 11 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT03497975/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT03497975/SAP_001.pdf